CLINICAL TRIAL: NCT05643040
Title: Comparison of Perioperative Analgesic Efficacy in Patients Who Had Femoral Nerve Block, Adductor Canal Block and 4in1 Block Applied in Knee Surgery
Brief Title: Comparison of Perioperative Analgesic Efficacy of Femoral Nerve Block, Adductor Canal Block and 4in1 Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Funda Atar, Diskapi Yildirim Beyazit Education and Research Hospital, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 06/06/2022 139/13
Record Dates: First submitted 2022-11-23; First posted 2022-12-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Block; Analgesia
Keywords: 4 in 1 block; femoral block; adductor canal block
MeSH Terms: conditions — Bites and Stings; Agnosia

STUDY DESIGN:
Intervention Model Description: Group I: Femoral nerve block Group II: Adductor canal block Group III: 4in1 block
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- femoral nerve block (Experimental): To evaluate the intraoperative analgesia effectiveness of femoral nerve block in patients who will have knee surgery.
  Interventions: Other: femoral nerve block
- adductor canal block (Experimental): To evaluate the intraoperative analgesia effectiveness of adductor canal block in patients who will have knee surgery.
  Interventions: Other: adductor canal block
- 4in1 block (Experimental): To evaluate the intraoperative analgesia effectiveness of 4in1 block in patients who will have knee surgery.
  Interventions: Other: 4in1 block

INTERVENTIONS:
Other: femoral nerve block — To evaluate the intraoperative analgesia effectiveness of femoral block in patients who will have knee surgery.
  Arms: femoral nerve block
Other: adductor canal block — To evaluate the intraoperative analgesia effectiveness of adductor canal block in patients who will have knee surgery.
  Arms: adductor canal block
Other: 4in1 block — To evaluate the intraoperative analgesia effectiveness of 4in1 block in patients who will have knee surgery.
  Arms: 4in1 block

SUMMARY:
Central neuraxial and regional anesthesia and analgesia techniques significantly reduce perioperative morbidity and mortality in the knee and below-knee surgeries.Nerve blocks appear to have better analgesic efficacy compared to placebo or patient-controlled analgesia (PCA). In addition, opioid-related side effects such as postoperative nausea, vomiting, pruritus, sedation, and respiratory depression are less. Therefore, interest in regional blocks such as femoral, sciatic, adductor, combined femoral, and sciatic is increasing. The knee joint is innervated by various nerves (genicular nerves) from the femoral, obturator, and sciatic nerves, and a comprehensive but simple technique is needed for postoperative analgesia. Complete and comprehensive postoperative analgesia was possible with this block, a simple single injection technique. The aim of our study is to evaluate the intraoperative analgesia efficacy of femoral, adductor canal block, and 4in1 block in patients who will undergo knee surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of >18
* undergone knee surgery
* American Society of Anesthesiologists (ASA) classification I-III group.

Exclusion Criteria:

* Patients who do not want to participate in the study coagulopathy peripheral neuropathy local anesthetic drug allergy chronic opioid users anticoagulant users pregnant patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
intraoperative analgesia efficacy | perioperative period
  The aim of our study is to evaluate the intraoperative analgesia efficacy of femoral, adductor canal block and 4in1 block in patients who will undergo knee surgery.

SECONDARY OUTCOMES:
postoperative analgesia efficacy | perioperative period
  The aim of our study is to evaluate the postoperative analgesia efficacy of femoral, adductor canal block and 4in1 block in patients who will undergo knee surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Science, Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodgers A, Walker N, Schug S, McKee A, Kehlet H, van Zundert A, Sage D, Futter M, Saville G, Clark T, MacMahon S. Reduction of postoperative mortality and morbidity with epidural or spinal anaesthesia: results from overview of randomised trials. BMJ. 2000 Dec 16;321(7275):1493. doi: 10.1136/bmj.321.7275.1493. PMID 11118174
- [Background] Roy R, Agarwal G, Pradhan C, Kuanar D. Total postoperative analgesia for total knee arthroplasty: Ultrasound guided single injection modified 4 in 1 block. J Anaesthesiol Clin Pharmacol. 2020 Apr-Jun;36(2):261-264. doi: 10.4103/joacp.JOACP_260_19. Epub 2020 Jun 15. PMID 33013045